CLINICAL TRIAL: NCT00006142
Title: Study of a Phenylalanine Restricted Diet During Pregnancy to Prevent Symptoms in Offspring of Patients With Phenylketonuria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Texas (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Prevention
Other Study IDs: 199/15326; UTMB-83-188
Record Dates: First submitted 2000-08-03; First posted 2000-08-04 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-08

CONDITIONS: Phenylketonuria
Keywords: inborn errors of metabolism; phenylketonuria; rare disease
MeSH Terms: conditions — Phenylketonurias; Metabolism, Inborn Errors; Rare Diseases

INTERVENTIONS:
Behavioral: phenylalanine restricted diet

SUMMARY:
OBJECTIVES:

I. Assess the impact of a phenylalanine restricted diet during pregnancy on symptoms in offspring of patients with phenylketonuria.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a multicenter study.

Patients receive a phenylalanine restricted diet based on a medical food such as Phenyl-free, Lofenalac, PKU 3, or Maximum XP (may be supplemented with tyrosine as needed) to achieve a target blood phenylalanine level of 2-6 mg/dL. The diet begins approximately 3 months prior to conception and continues until delivery of the baby. Patients are evaluated once a month before conception and weekly during pregnancy. Patients also undergo sonographic examination at 8, 20, 28, and 34 weeks gestation. At birth, the cord blood is evaluated for plasma amino acids. If the baby is found to have an elevated phenylalanine level, blood and urine are obtained to determine the baby's genetic status. Phenylalanine and tyrosine levels are checked in the baby daily for three days after birth.

The baby is followed for physical and mental development at 3 and 6 months and then annually thereafter.

ELIGIBILITY:
* Women with diagnosis of phenylketonuria who are planning on becoming pregnant Slightly elevated phenylalanine level (hyperphe variant) allowed

Min Age: 0 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1983-12

CONTACTS AND LOCATIONS:
Overall Officials: Bobbye M. Rouse, Study Chair — University of Texas